#### **Research Consent Form**

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates



OHRS Version: 1.31.2020

**Protocol Title:** PREPARE: PRevention using EPA against coloREctal cancer

**DF/HCC Principal Investigator(s) / Institution(s):** Dr. Andrew Chan, MPH /

Massachusetts General Hospital

**Main Consent** 

### INTRODUCTION AND KEY INFORMATION

All research is voluntary. It is your choice whether you take part in this research or not. If you decide to participate, please sign and date at the end of this form. We will give you a copy and you can refer to this consent form at any time.

The following is a short summary of this research study to help you decide whether you would like to be a part of this study. More detailed information is provided later in this form.

For purposes of this research, you will be referred to as a "participant."

### 1. Why am I being invited to take part in a research study?

You are invited to take part in this research study, because you have previously undergone a colonoscopy at Massachusetts General Hospital and had an adenoma removed during this previous procedure.

### 2. Why is this research being done?

This research study is studying a drug intervention as a possible chemoprevention strategy for colorectal cancer.

## 3. Who is supporting this research?

The National Cancer Institute (NCI) of the National Institutes of Health (NIH) is supporting this research study by providing funding for this research study.


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | ] |
|---|---|---|
| Research Consent Form | | |
| Dana-Farber/ Harvard Cancer Center | | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners N | etwork Affiliates | OHRS Version: 1 31 2020 |

### 4. What does this research study involve and how long will it last?

This research study involves intervention of AMR101 (VASCEPA) regimen (4 g/day) for 8-12 weeks with two study visits, including one prior to intervention and the other one after completion of the intervention.

The names of the study drug involved in this study are/is:

A daily AMR101 (VASCEPA).

AMR101 (icosapent ethyl) is a prescription medicine for adults to lower blood levels of triglycerides. It is supplied as a liquid-filled gel capsule for oral administration. The standard dose is 4 grams per day (administered as 8 half-gram capsules). Each 0.5-gram capsule of AMR101 contains 0.5 gram of icosapent ethyl, which is an ethyl ester of the omega-3 fatty acid eicosapentaenoic acid (EPA). EPA possesses triglyceride-lowering and anti-inflammatory activities and has been suggested to be beneficial for a variety of health outcomes in adults, including coronary heart disease, stroke, type 2 diabetes, depression, and inflammatory bowel disease, although the data are not univocal. Increasing evidence supports the anticancer effect of EPA.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits during which you will undergo a flexible sigmoidoscopy procedure, provide a blood draw, a urine sample, and complete a lifestyle questionnaire and a nutritional survey. Up to 24 mucosal biopsies will be taken, and a rectal brushing and stool specimen will also be collected.

You will receive study treatment of AMR101 for a minimum of 8 weeks and will be followed for a maximum of 12 weeks.

It is expected that about 80 people will take part in this research study.

Information about you and your health is personal and private. Generally, it cannot be obtained without your written permission. By signing this form, you are providing that permission and your information may be obtained and used in


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | |
|---|---|---|
| Research Consent Form | | |
| Dana-Farber/ Harvard Cancer Center | | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners N | etwork Affiliates | OHRS Version: 1.31,2020 |

accordance with this informed consent and as required or allowed by law. This means that researchers may obtain information regarding your past medical history, as well as specimens and samples from previous health care providers such as hospitals and labs.

### 5. What are the risks to participating in this study?

There are risks to taking part in any research study. We want to make sure you know about a few key risks right now. There may also be rare, serious and potentially life-threatening side effects. More detailed information is provided in the "What are the risks or discomforts of the research study?" section.

There is a risk that you could have side effects from the AMR101 drug.

Some of the most common side effects associated with participating in the study that doctors know about are:

- Arthralgia (or joint stiffness) associated with AMR101 treatment
- Dental pain and pain in the throat
- Mild to moderate gastrointestinal effects that include stomach pain, nausea, loss of appetite, constipation, or diarrhea.
- Perforation (or a hole) in the intestinal wall associated with flexible Sigmoidoscopy

## 6. Will being in this study benefit me in any way?

We do not know if taking part in this study will benefit you. This study may help researchers learn information that could help people in the future.

### 7. What are my options?

Instead of being in this research study, you have other options which may include the following:

- Receive standard treatment including follow-up colonoscopy at the appropriate surveillance interval as prescribed by your physician.
- Receive the same drugs, but not as part of a research study.
- Decide not to participate in this research study 

| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | ] |
|---|---|---|
| Research Consent Form | | ] |
| Dana-Farber/ Harvard Cancer Center | | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners N | etwork Affiliates | OHRS Version: 1.31.2020 |

• Participate in another research study.

If you choose not to participate, are not eligible to participate, or withdraw from this research study, this will not affect your present or future care and will not cause any penalty or loss of benefits to which you are otherwise entitled.

We encourage you to take some time to think this over, to discuss it with other people and your primary doctor, and to ask questions at any time.


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |



### A. WHY IS THIS RESEARCH STUDY BEING DONE?

This research study is a chemoprevention clinical trial, designed tests the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved AMR101 as a treatment for any disease.

In this research study, we are investigating the use of AMR101 as a potential chemopreventive agent to reduce risk of colorectal cancer. AMR101 is made of marine omega-3 fatty acid, which is a family of natural substances found in the oil of certain fish, such as salmon and mackerel. Marine omega-3 fatty acid cannot be produced in sufficient amount by our human body and has to be obtained through diet or supplemented to maintain normal function of our body.

Marine omega-3 fatty acid is well known to reduce inflammation. Substantial evidence has demonstrated that people with higher intake of marine omega-3 fatty acid have a lower likelihood of developing colon cancer. However, there remains uncertainty surrounding this mode of action.

By performing this research study, we hope to investigate the mode of action of marine omega-3 fatty acid on the gut bacteria and the immune system, which may lead to the use of marine omega-3 fatty acid as an effective agent to prevent colon cancer.

### B. WHAT IS INVOLVED IN THE RESEARCH STUDY?

You will be given a study medication (AMR101) for the duration of the study (8-12 weeks).

## Before the research starts (screening):

After signing this consent form, you will be asked to undergo some screening tests or procedures to find out if you can be in the research study. Many of these tests and procedures are likely to be part of regular care and may be done even if it turns out that you do not take part in the research study. If you have had


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | |
|---|---|---|
| Research Consent Form | | |
| Dana-Farber/ Harvard Cancer Center RIDMC/RCH/RWH/DECI/MGH/Partners I | Notwork Affiliatos | OHPS Version: 1 31 2020 |

some of these tests or procedures recently, they may or may not have to be repeated.

- A medical history, which includes questions about your health, current medications, and any allergies.
- **Performance status**, which evaluates how you are able to carry on with your usual activities.

If these tests show that you are eligible to participate in the research study, you may begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

### **Study Treatment Overview:**

Oral Study Drug(s): Each study treatment cycle lasts 8 weeks during
which time you will be taking the study drug 2 times per day unless dose
reduction is indicated. This will continue for up to 12 weeks.

If you take part in this research study, you will be given a drug diary. You will be asked to document information in the drug diary about the study treatment you are being asked to take.

### Study Visit: Initial (baseline) Visit

At the baseline visit, your physician will obtain written, informed consent for the study as well as a standard clinical consent to perform a flexible sigmoidoscopy. This flexible sigmoidoscopy is similar to your previous colonoscopy. During the procedure the endoscope is only inserted a few inches past your rectum. This flexible sigmoidoscopy will be performed without a bowel preparation, which means that you do not have to drink any laxative preparation in advance of the procedure. At this visit, you will undergo measurements of height, weight, waist and hip circumference and provide blood and urine specimens. A study gastroenterologist will then perform the flexible sigmoidoscopy, advancing only about 6-10 inches. Thus, you will not require any sedation for this procedure. No more than a total of 24 mucosal biopsies will be taken from the rectum and sigmoid colon and immediately placed in collection tubes.

### This visit will involve the following:


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM |
|-----------------------|
| Bosserch Consont Form |

#### Research Consent Form

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

 Clinical Exams: During this visit you will have a physical exam and you will be asked questions about your general health and specific questions about any problems that you might be having and any medications you may be taking.

OHRS Version: 1.31.2020

- A lifestyle questionnaire and a nutritional survey. Our research assistant will help you complete a questionnaire and a nutritional survey which evaluate your lifestyle risk factors, current nutritional intake, and dietary trends.
- Blood samples drawn. Approximately 2.5 teaspoons of blood (12 mLs)
- Flexible sigmoidoscopy, where up to 24 normal colon tissue biopsies will be collected.
- Urine sample provided.
- Stool specimen collected (during flexible sigmoidoscopy)
- Confirm or schedule final visit, which will occur at least 8 weeks but no more than 12 weeks following this initial visit.

### Study Visit 2: Final Visit, study treatment ends

### This visit will involve the following:

- Return drug bottle with any remaining pills.
- Clinical exams: During this visit you will have a brief physical exam and you will be asked questions about your general health and specific questions about any problems that you might be having and any medications you may be taking.
- A second lifestyle questionnaire and a nutritional survey
- Blood samples drawn. Approximately 2.5 teaspoons of blood (12 mLs)
- Urine sample provided.
- Flexible sigmoidoscopy, where up to 24 normal colon tissue biopsies will be collected.
- Stool specimen collected (during flexible sigmoidoscopy)

### Research Study Plan:

| Visit 1 | Treatment<br>Period | Visit 2 |
|---------------|---------------------|-------------|
| Initial Visit | 1 CHOC | Final Visit |


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM |
|-------------------|

### Research Consent Form

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

| OHRS | version: | 1.31.2020 |
|------|----------|-----------|

| Medical History & Physical Exam | Х | | X |
|----------------------------------------------|---|---|---|
| Blood Draw | Х | | Х |
| Urine Collection | Х | | Х |
| Flexible Sigmoidoscopy | Х | | Х |
| Normal Colon Tissue Biopsy | Х | | Х |
| Complete | Х | | Х |
| Questionnaires and nutritional surveys | ^ | | ^ |
| Stool collection | X | | X |
| Receive study drug <sup>a</sup> | X | | |
| Take 8 capsules of the study drug per day | | X | |
| for a minimum of 8 and maximum of 12 | | | |
| weeks <sup>b</sup> | | | |
| Return pill bottle with unused drug capsules | | | X |

<sup>a: You will take 4 capsules of study drug twice daily (8 capsules per day) until your final visit 8-12 weeks after your initial visit.
b: Should you experience GI-related side effect(s) such as nausea.</sup> 

### Planned Follow-up:

We would like to keep track of your medical condition. Between the initial and final visits, a study coordinator will contact you weekly to make sure you aren't experiencing any adverse side effects and track your use of the study drug. After the study we will also contact you for one month to follow-up on additional information, including any use of fish oil supplements and results of any follow-up colonoscopies. After the study is completed, we may contact you with the contact information you provided for future related studies. Keeping in touch with you and checking your condition helps us look at the long-term effects of the research study.

In addition, you can stop participating in the research study at any time, however, the FDA requires that any information collected up to the point of your withdrawal cannot be removed from the study.

### **Collection and Processing of Biospecimens:**

Immediately following each flexible sigmoidoscopy, urine specimens will be aliquoted and blood specimens will be centrifuged into plasma and buffy coat. Stool specimens will be stored in a cryovial and immediately frozen. Colon


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

vomiting, constipation, diarrhea, inform the study team for potential study drug dose reduction to 4 capsules of study drug per day.



biopsies will be immediately frozen for future RNA-seq analysis. Yield from these procedures typically exceeds requirements for RNA-seq. Thus, any excess colon tissue will be banked for future studies. All aliquots of stool, urine, plasma, buffy coat, and tissue will be frozen at -80°C until analysis which will be conducted by a third party.

### C. WHAT ARE THE RISKS OR DISCOMFORTS OF THE RESEARCH STUDY?

There are risks to taking part in any research study. One risk is that you may get a study drug that does not help treat your disease or that makes your condition or disease worse. Another risk is that there may be side effects.

All cancer treatments can have side effects, which can range from mild and reversible to severe, long lasting and possibly life-threatening. There is a great deal of variability among side effects of different cancer treatments and between individuals. In a research study, all of the risks or side effects may not be known before you start the study. You need to tell your doctor or a member of the study team immediately if you experience any side effects.

Everyone in the research study will be watched carefully for side effects. You will be monitored during the administration of study drugs. If you experience side effects, they may go away after you stop taking the study drug. Some side effects can be mild; but others can be long lasting and may never go away. Some may be life-threatening or fatal.

Since the effect of the study drug(s) taken with other medications may not be known, it is important that you tell the research doctor about all prescription and non-prescription drugs, herbal preparations and nutritional supplements that you are taking or planning to take. There may also be some foods that you should avoid while on this research study and your research doctor will review this information with you.

During the research study, you will be notified of newly discovered side effects or significant findings, which may affect your health or willingness to participate. You may be asked to sign a new consent form that shows that you have been informed of new information relating to this research study.

### Risks Associated with AMR101 Use:


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | |
|---|---|---|
| Research Consent Form | | |
| Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners I | Network Affiliates | OHRS Version: 1.31.2020 |

#### Occasional

- Arthralgia (pain in a joint) is one of the most commonly reported adverse events with an occurrence rate of 2.3%.
- Dental pain and pain in the throat have also been reported.
- Mild to moderate gastrointestinal side effects that may include stomach pain, nausea, loss of appetite, constipation, or diarrhea.

Cancer research often includes biopsies, scans, x-rays that are also provided as routine care. The following describes the side effects of procedures done only for the purposes of research.

### Risks Associated with Flexible Sigmoidoscopy:

Flexible sigmoidoscopy is generally a safe test although rare complications can occur. These can include some mild pain or discomfort, like a feeling of fullness, felt during this test. Even more rarely (less than 1 in 10,000 times), a hole (perforation) can be made in the side of the rectum or colon that can require surgical intervention.

### **Risks Associated with Biopsies:**

Biopsies are normally performed under the guidance of an imaging technique. Each procedure requires a separate consent prior to the biopsy. Biopsies of the colon are performed by inserting biopsy forceps through the endoscope and removing a small piece of tissue. Minor bleeding or pain, the most common complications resulting from endoscopic biopsy, complicate less than 1 of every 3000 (0.03%) colonoscopic procedures. This study requires 24 biopsies per procedure. A study of the safety of research biopsies by the National Institutes of Health has determined that more than 20 biopsies per procedure, including as many as 85, is well tolerated and appears to have no more than minimal risk without increasing the risk of otherwise routine colonoscopy.

### The risks may include:

- Pain and discomfort. The amount of pain and discomfort will vary, depending on the location of the biopsy site. These risks can be discussed with the study doctor.
- Minor bleeding at the biopsy site. Major bleeding episodes that require blood transfusions or hospitalization are extremely rare.


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | |
|---|---|---|
| Research Consent Form | | |
| Dana-Farber/ Harvard Cancer Center | | |
| RIDMC/RCH/RWH/DECI/MGH/Partners No | etwork Affiliates | OHDS Version: 1 31 3030 |

- Tenderness at the biopsy site.
- Scarring at the biopsy site.
- Rarely, an infection at the biopsy site.

Uncommonly, complications from biopsies can be life threatening. As with any interventional procedure, other potentially serious complications from bleeding or organ damage may occur. These might require additional surgical intervention.

### **Risks Associated with Phlebotomy:**

You will have 2 blood draws during the study. A small amount of blood (12 mLs or approximately 2.5 teaspoons) will be taken at each blood draw and poses minimal risk. The total blood collected during the study will be 24 mLs. The risk of blood draws include:

- Discomfort at the site of blood draw.
- Bruising, bleeding, infection.
- Rarely fainting.

### **Reproductive Risks**:

The drugs used in this research study may affect a fetus.

While participating in this research study, you should not:

- become pregnant
- nurse a baby
- father a baby

We can provide counseling about preventing pregnancy for either male or female study participants. Let your doctor know immediately if you become pregnant or find out that you are going to be the father of a child.

If your partner becomes pregnant while you are on the study, it may be critical to share information regarding your participation in this research study with that person. Your research doctor should also be told if this happens.

### Risks of Tissue Collection for Biobanking:


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |



Generally, hospitals will keep some of your tissue. There is a small risk that when this tissue is collected and the sample is submitted to the biobank, your tissue could be used up and unavailable for use in the future.

### Non-Physical Risks:

Because of side effects or the time required for tests and clinic visits while you are on this research study, you may be unable to keep up with your normal daily activities.

The questionnaires used in this study may be upsetting. If you find the questionnaires upsetting, you may speak with the research doctor or ask to be referred for additional emotional support.

# D. WHAT WILL HAPPEN IF I AM REMOVED FROM THE STUDY OR DECIDE TO END MY PARTICIPATION IN THE RESEARCH?

You may be taken off the research study for any reason including:

- It is considered to be in your best interest
- The study treatment or procedures are found to be unsafe or ineffective
- There is any problem with following study treatments and procedures
- You are a female and become pregnant or plan to become pregnant
- Your condition worsens
- A decision is made to end the study
- Or for other unforeseen reasons that make it necessary to stop your participation in the research study

You can also choose to stop participating in the research study at any time. Tell the research doctor if you are thinking about stopping or decide to stop. He or she will tell you how to stop. Leaving the research study will not affect your medical care outside of the research study.

It is important to tell the research doctor if you are thinking about stopping so your research doctor can evaluate the risks from stopping the drug.

#### 

| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |



It is important to note that although you may withdraw from study participation, the FDA requires that any information collected up to the point of your withdrawal cannot be removed from study records. Additionally, the research doctor may consult public records after you have withdrawn from the study.

If you decide to withdraw from a study that involves de-identified samples, it will not be possible to remove the samples and data that have already been submitted to a database or biobank.

### E. WHAT ARE THE BENEFITS OF THIS RESEARCH STUDY?

Taking part in this research study may or may not benefit you. We hope the information learned from this research study will provide more information about the effect of daily 4-gram AMR101 treatment on fatty acid composition in colorectal tissue, on the gut microbiome and metabolome, and gene expression profile of colorectal tissue among individuals with a history of colorectal adenoma.

### F. WILL I BE PAID TO TAKE PART IN THIS RESEARCH STUDY?

You will be compensated for participating in this research study. Participants who complete the baseline visit and protocol will receive \$100.00 (US) compensation. Patients who complete the end visit and protocol will receive an additional \$100.00 (US) compensation. Additionally, if you require parking for your two study visits, you will receive up to four hours of parking at no charge to you.

We may use your samples and information to develop a new product or medical test to be sold. The sponsor and hospital may benefit if this happens. There are no plans to pay you if your samples are used for this purpose.

### G. WHAT ARE YOUR COSTS?

Taking part in this research study may lead to added costs to you or your insurance company. This may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your disease. You may:

Have more travel costs


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | |
|---|---|---|
| Research Consent Form | | |
| Dana-Farber/ Harvard Cancer Center | | |
| RIDMC/RCH/RWH/DECI/MGH/Partners No | etwork Affiliates | OHDS Version: 1 31 3030 |

- Need to take more time off work
- Have other additional personal costs

You will not be charged for the study drug (AMR101) or procedures.

You or your insurance company will be charged for portions of your care during this research study that are considered standard care. Standard of care is the care that you would receive regardless of whether you were enrolled in the study or not. You may be responsible for co-payments, co-insurance, premiums and deductibles that are typical for your insurance coverage. This includes the cost of tests, procedures, or medicines to manage any side effects, unless you are told that certain tests, done for research only, are supplied at no charge.

If you have questions about your insurance coverage, or the items you might be required to pay for, please call financial services for information. The contact information for financial services are:

Massachusetts General Hospital: (617) 726-2191

The National Cancer Institute provides an online resource to help people participating in cancer clinical trials understand which services their insurance company is required by law to pay. This can be found at the website below or can be provided by the study team:

<u>www.cancer.gov</u> or 1-800-4-CANCER (1-800-422-6237)

# H. WHAT HAPPENS IF I AM INJURED OR BECOME SICK BECAUSE I TOOK PART IN THIS RESEARCH STUDY?

If you think you have been injured as a result of taking part in this research study, tell the person in charge of this research study as soon as possible. The research doctor's name and phone number are listed in this consent form.

#### 

| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |



BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates OHRS Version: 1.31.2020

The treating hospital will offer you the care needed to treat injuries directly resulting from taking part in this research. These treatments may be billed to you or your insurance company. You will be responsible for deductibles, co-payments and co-insurance. There are no plans to pay you or give you other compensation for the injury.

You do not give up your legal rights by signing this form.

We will need to collect certain personal information about you for insurance or payment reporting purposes, such as your name, date of birth, gender, social security number or Medicare identification number and information related to this research study. We may be required to report this information to the Centers for Medicare & Medicaid Services. We will not use this information for any other purpose.

If you go to the Emergency Room or to another hospital or doctor it is important that you tell them that you are in this research. If possible, you should give them a copy of this consent form.

### I. WHOM DO I CONTACT IF I HAVE QUESTIONS ABOUT THE RESEARCH STUDY?

If you have questions about the study, please contact the research doctor or study staff as listed below:

Massachusetts General Hospital

- Andrew T. Chan, MD, MPH: (617) 726-3212
- Mingyang Song, MD, ScD: (617) 643-4464
- Marina Magicheva-Gupta, MPH: (617) 726-4807

## 24-Hour Contact: Massachusetts General Hospital, Andrew Chan, MD at (617) 726-7777, pager 31100.

For questions about your rights as a research participant, please contact a representative of the Office for Human Research Studies at Dana-Farber Cancer Institute (617) 632-3029. This can include questions about your participation in the study, concerns about the study, a research related injury, or if you feel/felt under pressure to enroll in this research study or to continue to participate in this research study.


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |



### J. RETURN OF RESEARCH RESULTS

Tests done on samples in this research study are only for research and have no clear meaning for your health care. For this reason, your study doctor will not share the results with you.

### K. CLINICALTRIALS.GOV (CT.GOV)

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This web site will not include information that can identify you. At most, the web site will include a summary of the results. You can search this web site at any time.

### L. FUTURE USE OF DATA AND SPECIMENS

Your personal information and/or biospecimens collected during this study may be stored and used for future research. Any personal identifiers will be removed, before they are shared, so that the information or samples cannot be linked back to you. As a result, we will no longer be able to identify and destroy them.

Investigators, including investigators from collaborating institutions, can request this data and samples for new research. Samples and data may also be shared with outside non-profit academic investigators as well as with for-profit pharmaceutical investigators or commercial entities, with whom we collaborate.

You will not be asked to provide additional informed consent for the use of your de-identified information or samples in future research.

Future research studies may include genetic research. Your genes are unique to you. At this time, you cannot be identified through this research, if the samples and specimens are de-identified. There is a risk that you might be reidentified in the future as genetic research progresses


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |



### M. CONFIDENTIALITY

We will take measures to protect the privacy and security of all your personal information, but we cannot guarantee complete confidentiality of study data.

Medical information created by this research study may become part of your hospital medical record and may be forwarded to your primary doctor. Information that does not become part of your medical record will be stored in your study file. It may also become part of a research database.

Participation in this study involves providing a specimen of your tissue; please know that if the research doctor leaves the institution, the research and the tissue might remain at the research doctor's current institute or might be transferred to another institution.

The study team plans to publish the results of this research study and when we do, we may be asked to make the data we collect available to other researchers. We will not include information that identifies you in any publications or to the researchers who request the data to do additional research.

Your de-dentified specimens or genetic data may also be placed into one or more publicly-accessible scientific databases. Through such databases, researchers from around the world will have access to de-identified samples or data for future research.

There is a risk that de-identified research data that is shared with outside collaborators may be reidentified. When de-identified data and specimens are shared with outside collaborators agreements limit what the outside collaborators can do with the information to help prevent reidentification.

### N. FINANCIAL DISCLOSURES

It is possible that certain researchers on this study may have earned money from, or own some publicly-traded stock in, the company that makes or is developing the study drug. The amount of money that a researcher may earn and still take part in research is limited by the Harvard Medical School Faculty of Medicine Policy on Conflicts of Interest and Commitment. If you have further questions, please speak with a member of the study team or contact the Dana-


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |



Farber Cancer Institute Office of Research Integrity at 617-432-4557 or researchintegrity@dfci.harvard.edu.

### O. CERTIFICATE OF CONFIDENTIALITY (COC)

To help protect your privacy, we have been issued a Confidentiality Certificate from the National Institutes of Health (NIH). With this Certificate, the researchers on this study cannot be forced (for example, by court subpoena) to disclose information that may identify you in federal, state, or local civil, criminal, administrative, legislative or other proceedings.

Disclosure will be necessary upon request of a United States federal or state government agency sponsoring the project that will be used for audit or program evaluation purposes or to meet the requirements of the federal Food and Drug Administration (FDA).

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family or even the research doctor from voluntarily releasing information about yourself or your involvement in this research. If an insurer, medical care provider, or employer learns about your participation, and obtains your consent to receive research information, then we cannot use the Certificate of Confidentiality to withhold this information. This means that you and your family must actively protect your own privacy.

The Certificate of Confidentiality cannot be used to prevent disclosure to state or local authorities when there is a duty to report concerns of abuse, neglect, selfharm or a danger to others.

## P. GENETIC RESEARCH

This research will involve genomic and germline testing.

The Genetic Information Nondiscrimination Act of 2008 (GINA) is a federal law that protects Americans from being treated unfairly because of differences in their DNA that may affect their health, and may prevent discrimination by health insurers and employers based on genetic information. GINA is intended to ease concerns about discrimination that might keep some people from getting genetic tests that could benefit their health and enable people to take part in research 

| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |



studies such as this without fear that their DNA information might be used against them by health insurers or their workplace. This protection does not extend to disability or life insurance. Additional information can be found at <a href="http://www.genome.gov/10002328">http://www.genome.gov/10002328</a>.

As part of this study, your de-identified specimens or genetic data may be placed into one or more publicly-accessible scientific databases, such as the National Institutes of Health's Database for Genotypes and Phenotypes (dbGaP). Through such databases, researchers from around the world will have access to de-identified samples or data for future research.

### Q. PRIVACY OF PROTECTED HEALTH INFORMATION (HIPAA AUTHORIZATION)

The Health Insurance Portability and Accountability Act (HIPAA) is a federal law that requires Dana-Farber/Harvard Cancer Center (DF/HCC) and its affiliated research doctors, health care providers, and physician network to protect the privacy of information that identifies you and relates to your past, present, and future physical and mental health conditions ("protected health information"). If you enroll in this research study, your "protected health information" will be used and shared with others as explained below.

# 1. What protected health information about me will be used or shared with others during this research?

- Existing medical records, including mental health records.
- New health information created from study-related tests, procedures, visits, and/or questionnaires

### 2. Why will protected information about me be used or shared with others?

The main reasons include the following:

- To conduct and oversee the research described earlier in this form;
- To ensure the research meets legal, institutional, and accreditation requirements;
- To conduct public health activities (including reporting of adverse events or situations where you or others may be at risk of harm); and

#### 

| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | ] |
|---|---|---|
| Research Consent Form | | |
| Dana-Farber/ Harvard Cancer Center | | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners N | etwork Affiliates | OHRS Version: 1.31.2020 |

• To provide the study sponsor with information arising from an adverse event or other event that relates to the safety or toxicity of the drug(s) used in the study and for the purpose of this or other research relating the

- To better understand the diseases being studied and to improve the design of future studies; and,
- Other reasons may include for treatment, payment, or health care operations. For example, some medical information produced by this research study may become part of your hospital medical record because the information may be necessary for your medical care. (You will also be given a notice for use and sharing of protected health information.)

### 3. Who will use or share protected health information about me?

study drug(s) and their use in cancer;

 DF/HCC and its affiliated research doctors and entities participating in the research will use and share your protected health information. In addition, other DF/HCC offices that deal with research oversight, billing or quality assurance will be able to use and share your protected health information.

## 4. With whom outside of DF/HCC may my protected health information be shared?

While all reasonable efforts will be made to protect the confidentiality of your protected health information, it may also be shared with the following entities:

- Outside individuals or entities that have a need to access this information
  to perform functions relating to the conduct of this research such as
  analysis by outside laboratories on behalf of DF/HCC and its affiliates (for
  example, data storage companies, insurers, or legal advisors).
- The sponsor(s) of the study, its subcontractors, representatives, business partners, and its agent(s): Cancer Institute and the National Institutes of Health.
- Other research doctors and medical centers participating in this research, if applicable
- Federal and state agencies (for example, the Department of Health and Human Services, the Food and Drug Administration, the National Institutes of Health, and/or the Office for Human Research Protections), or


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | ] |
|---|---|---|
| Research Consent Form | | ] |
| Dana-Farber/ Harvard Cancer Center | atural ACCU | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners N | etwork Affiliates | OHRS Version: 1.31.202 |

other domestic or foreign government bodies if required by law and/or necessary for oversight purposes. A qualified representative of the FDA and the National Cancer Institute may review your medical records.

- Hospital accrediting agencies
- A data safety monitoring board organized to oversee this research, if applicable

Some who may receive your protected health information may not have to satisfy the privacy rules and requirements. They, in fact, may share your information with others without your permission.

## 5. For how long will protected health information about me be used or shared with others?

 There is no scheduled date at which your protected health information that is being used or shared for this research will be destroyed, because research is an ongoing process.

### 6. Statement of privacy rights:

- You have the right to withdraw your permission for the research doctors and participating DF/HCC entities to use or share your protected health information. We will not be able to withdraw all the information that already has been used or shared with others to carry out related activities such as oversight, or that is needed to ensure quality of the study. To withdraw your permission, you must do so in writing by contacting the researcher listed above in the section: "Whom do I contact if I have questions about the research study?"
- You have the right to request access to your protected health information that is used or shared during this research and that is related to your treatment or payment for your treatment, but you may access this information only after the study is completed. To request this information, please contact the researcher listed above in the section: "Whom do I contact if I have guestions about the research study?"

### 

| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | |
|---|---|---|
| Research Consent Form Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners | Network Affiliates | OHRS Version: 1.31.2020 |
| <ul><li>participating in this study</li><li>I have had all of my que</li><li>I am willing to participate</li></ul> | to read the consent and think<br>ly;<br>estions answered to my satisfa | action; |
| Signature of Participant or Legally Authorized Representat | Date<br>tive | |

Relationship of Legally Authorized Representative to Participant

## 

| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM |
|-------------------|

## **Research Consent Form**

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS Version: 1.31.2020

| To be completed by person obtaining consent: |
|---|
| Adult Participant |
| The consent discussion was initiated on (date). |
| Signature of individual obtaining consent: |
| Printed name of above: |
| Date: |
| A copy of this signed consent form will be given to the participant or legally authorized representative. |
| 1) The participant is an adult and provided consent to participate. |
| 1a) Participant (or legally authorized representative) is a non-English speaker and signed the translated Short Form in lieu of English consent document: |
| As someone who understands both English and the language used by the participant, I interpreted and/or witnessed, in the participant's language, the researcher's presentation of the English consent form. The participant was given the opportunity to ask questions. |
| Signature of Interpreter/Witness: |
| Printed Name of Interpreter/Witness: |
| Date: |
| ☐ 1b) Participant is physically unable to sign the consent form because: |
| ☐ The participant is illiterate. |
| ☐ The participant has a physical disability. |
| Other (please describe): |
| The consent form was presented to the participant who was given the opportunity to ask questions and who communicated agreement to participate in the research. |
| Signature of Witness: |
| Printed Name of Witness: |
| Date: |


| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |

| 1/6/2022 12:06 PM | | ] |
|---|---|---|
| Research Consent Form Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates OHRS Version: 1.31.2020 | | |
| The participant is an adult who lacks capacity to provide consent and his/her legally authorized representative: | | |
| <ul><li>2a) gave permission for the ac</li><li>2b) did not give permission fo</li></ul> | dult participant to participate r the adult participant to participate | |

## 

| DFCI Protocol Number: 19-402 | Approved Date (DFCI IRB Approval): 12/28/2021 |
|---|---|
| Date Posted for Use: 12/29/2021 | |